CLINICAL TRIAL: NCT06466551
Title: The Effect of Virtual Reality Goggles and Stress Ball Used During Intravenous Catheterization on Pain and Fear in Children: A Randomized Experimental Study
Brief Title: Effect of Virtual Reality Goggles and Stress Ball Use on Pain and Fear During IV Catheterization in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Didem Polat Kulcu, Assist. Prof. Dr., Toros University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Toros
Record Dates: First submitted 2024-06-03; First posted 2024-06-20 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pain, Procedural; Anxiety; Pain Management
Keywords: distraction; fear; pain
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders; Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Goggles Group (Experimental): Children in this group watched cartoons using virtual reality goggles starting 3 minutes before intravenous catheterization. Pain and fear were assessed before, during, and after the procedure.
  Interventions: Other: intravenous catheterization
- Stress Ball Group (Experimental): Children in this group used a stress ball as a distraction method starting 3 minutes before intravenous catheterization. Pain and fear were assessed before, during, and after the procedure.
  Interventions: Other: intravenous catheterization

INTERVENTIONS:
Other: intravenous catheterization — This randomized experimental study was planned to examine the effect of virtual reality goggles and squeezing a stress ball as a distraction method during intravenous catheter application on pain and fear in children aged 6-12 years.

SUMMARY:
Although distraction methods such as virtual reality glasses, watching videos, watching cartoons, etc. have been reported to reduce pain in the literature, studies on which method is more effective in reducing pain are limited. Considering the developmental period characteristics, virtual reality glasses and stress ball squeezing may be effective in the 6-12 age group during painful intervention. However, no study has been found in the literature on which technique is more effective (9-23). Therefore, investigating the effects of virtual reality goggles and stress ball squeezing on pain and fear in children aged 6-12 years as a distraction method during intravenous catheterization may enable nurses to determine the technique with high clinical usefulness in pain management.

DETAILED DESCRIPTION:
Provide a brief summary of the study, including the purpose, objectives, and brief methodology.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years
* Admitted to the pediatric unit of the hospital between June 20, 2024, and April 20, 2025
* Scheduled to undergo intravenous catheterization
* Having parental consent through a signed informed consent form
* Absence of mental or developmental retardation

Exclusion Criteria:

- Children for whom the first attempt at intravenous catheterization was unsuccessful

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores Assessed by the Wong-Baker FACES Pain Rating Scale | Baseline (before the procedure), Mid-procedure (during the procedure), Post-procedure (immediately after the procedure)
  Pain scores will be measured using the Wong-Baker FACES Pain Rating Scale. Scores will be recorded before, during, and after intravenous catheterization. Pain will be assessed immediately before the procedure (baseline), during the procedure (mid-procedure), and immediately after the procedure (post-procedure). Pain will be evaluated independently by the child (self-report), parent (observational), and researcher (observational).
Change in Fear Scores Assessed by the Children's Fear Scale | Baseline (before the procedure), Mid-procedure (during the procedure), Post-procedure (immediately after the procedure)
  Fear levels will be assessed using the Children's Fear Scale. Scores will be recorded before, during, and after intravenous catheterization. Fear will be assessed immediately before the procedure (baseline), during the procedure (mid-procedure), and immediately after the procedure (post-procedure). Fear will be evaluated independently by the child (self-report), parent (observational), and researcher (observational).

CONTACTS AND LOCATIONS:
Overall Officials: Didem Polat Külcü, Dr., Principal Investigator — Toros University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Toros Üniversty, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared for secondary research purposes upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available within 6 months after publication of the main study results and will be accessible for up to 3 years.
Access Criteria: Researchers must submit a methodologically sound proposal approved by an ethics committee. Data will be shared through secure, password-protected file transfer after signing a data use agreement.